CLINICAL TRIAL: NCT01355536
Title: Metabolic and Endocrine Status in Women With Prior Preterm Birth. A Cross Sectional, Case- Control Study
Brief Title: Metabolic and Endocrine Status in Women With Prior Preterm Birth
Status: Completed | Type: Observational
Sponsor: Namsos Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); The Royal Norwegian Ministry of Health (Other)
Responsible Party: Tina Eilertsen, MD, Hospital of Namsos
Other Study IDs: 46011600-57
Record Dates: First submitted 2011-05-09; First posted 2011-05-18 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Polycystic Ovary Syndrome; Preterm Birth; Diabetes Mellitus
Keywords: Preterm birth; Preterm labour; Polycystic Ovary Syndrome; PCOS; Diabetes Mellitus; Hyperandrogenism; Hirsutism; Ovarian cysts; Anti Muller Hormone; Hypertension
MeSH Terms: conditions — Polycystic Ovary Syndrome; Premature Birth; Diabetes Mellitus; Obstetric Labor, Premature; Hyperandrogenism; Hirsutism; Ovarian Cysts; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum,endometrial biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preterm birth group: Women with prior preterm birth
- Term birth group: Women with prior term birth

SUMMARY:
The prevalence of preterm birth is rising in most western countries. The causes of preterm birth is not fully understood and seem to be multifactorial. The endocrine and metabolic aspects are scarcely investigated.The main purpose of this study is to test the hypothesis that endocrine and metabolic factors associate to preterm births.

ELIGIBILITY:
Inclusion Criteria:

* One or more preterm birth in the given period of time
* Having Namsos Hospital as their local Hospital during pregnancy

Exclusion Criteria:

* Moved from the region of Mid- Norway at the time of the study
* Lack of communication skills in Norwegian or English
* Ongoing pregnancy
* Ongoing breastfeeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women in municipalities having Namsos Hospital as their local Hospital and with preterm births from January 1999 to Descember 2006 were identifed by searching birth protocols. These women were invited to participate in the preterm birth study group. As controls we identified the first term birth occuring in time after each preterm birth. These women were invited to participate in the term birth study group.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The prevalence of PCOS | one week after enrollment.
  The prevalence of PCOS will be assessed in both study groups and the difference between the groups will be reported.
The prevalence of Diabetes Mellitus | one week after enrollment
  The prevalence of Diabetes Mellitus will be assessed in both study groups and the difference between the groups will be reported.

SECONDARY OUTCOMES:
Ovarian antral follicle count | three years.
  Difference between study groups.
Difference in quality of life between study groups. | four years
  Quality of life will be assessed by using Short form 36 Health Survey Questionnaire (SF- 36)
Serum levels of androgens | one year
  Difference between study groups
Difference in anxiety between study groups. | four years
  Anxiety will be assessed by using Spielberger State Anxiety Inventory Y1 and Y2 (STAI Y1 and Y2).
Serum levels of AMH | One year
  Difference between study groups
Serum levels of glucose | One year
  Difference between study groups
Serum levels of insulin | One year
  Difference between study groups

CONTACTS AND LOCATIONS:
Overall Officials: Tina Eilertsen, MD, Principal Investigator — Namsos Hospital, Nord- Trøndelag Hospital Trust
Locations (1):
- Namsos Hospital, Nord- Trøndelag Hospital Trust, Namsos, Nord- Trøndelag, Norway

REFERENCES:
- [Derived] Eilertsen TB, Vanky E, Carlsen SM. Anti-Mullerian hormone in the diagnosis of polycystic ovary syndrome: can morphologic description be replaced? Hum Reprod. 2012 Aug;27(8):2494-502. doi: 10.1093/humrep/des213. Epub 2012 Jun 12. PMID 22693172
- [Derived] Eilertsen TB, Vanky E, Carlsen SM. Increased prevalence of diabetes and polycystic ovary syndrome in women with a history of preterm birth: a case-control study. BJOG. 2012 Feb;119(3):266-75. doi: 10.1111/j.1471-0528.2011.03206.x. Epub 2011 Dec 13. PMID 22168920